CLINICAL TRIAL: NCT01534273
Title: Single- and Multiple-Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of LY2886721 in Healthy Subjects
Brief Title: A Study of LY2886721 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14464; I4O-MC-BACJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers
Keywords: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — N-(3-(2-amino-4a,5,7,7a-tetrahydro-4H-furo(3,4-d)(1,3)thiazin-7a-yl)-4-fluorophenyl)-5-fluoropicolinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Single oral dose and/or once daily (QD) oral dosing for 14 consecutive days
  Interventions: Drug: Placebo
- 35 mg LY2886721 (Experimental): QD oral dosing for 14 consecutive days
  Interventions: Drug: LY2886721
- 70 mg LY2886721 (Experimental): Single oral dose or single oral dose followed by QD oral dosing for 14 consecutive days
  Interventions: Drug: LY2886721
- 140 mg LY2886721 (Experimental): Single oral dose
  Interventions: Drug: LY2886721

INTERVENTIONS:
Drug: LY2886721 — Administered orally.
  Arms: 140 mg LY2886721; 35 mg LY2886721; 70 mg LY2886721
Drug: Placebo — Administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this phase I study in healthy participants will be to evaluate the safety and tolerability of LY2886721 single and multiple doses, to evaluate how the body handles the drug, and to evaluate the drug's effect on the body.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and non-childbearing potential women
* Body mass index (BMI) between 18.0 and 32.0 kilograms per square meter (kg/m^2)
* Are reliable and willing to make yourself available for the duration of the study and are willing to follow study procedures and research unit policies

Exclusion Criteria:

* Taking over-the-counter or prescription medication with the exception of vitamins or minerals
* Smoke more than 10 cigarettes per day
* Drink more than 5 cups of caffeine containing beverages (for example, coffee, tea) per day

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Cohort A): Placebo: once daily (QD) oral dosing for 14 consecutive days
- 35 mg LY2886721 (Cohort A): 35 milligrams (mg) LY2886721: QD oral dosing for 14 consecutive days
- Placebo (Cohort B): Placebo: single oral dose (Period 1) followed by QD oral dosing for 14 consecutive days (Period 2)
- 70 mg LY2886721 (Cohort B): 70 mg LY2886721: single oral dose (Period 1) followed by QD oral dosing for 14 consecutive days (Period 2)
- Placebo (Cohort C): Placebo: single oral dose
- 70 mg LY2886721 (Cohort C): 70 mg LY2886721: single oral dose
- 140 mg LY2886721 (Cohort C): 140 mg LY2886721: single oral dose
Period: Period 1
Arm/Group | Placebo (Cohort A) | 35 mg LY2886721 (Cohort A) | Placebo (Cohort B) | 70 mg LY2886721 (Cohort B) | Placebo (Cohort C) | 70 mg LY2886721 (Cohort C) | 140 mg LY2886721 (Cohort C)
Started | 3 | 6 | 2 | 7 | 3 | 3 | 6
Received at Least 1 Dose of Study Drug | 3 | 6 | 2 | 7 | 3 | 3 | 6
Completed | 3 | 6 | 2 | 6 | 3 | 3 | 6
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Period 2
Arm/Group | Placebo (Cohort A) | 35 mg LY2886721 (Cohort A) | Placebo (Cohort B) | 70 mg LY2886721 (Cohort B) | Placebo (Cohort C) | 70 mg LY2886721 (Cohort C) | 140 mg LY2886721 (Cohort C)
Started | 0 (Participants in Cohort A participated in only 1 treatment period.) | 0 (Participants in Cohort A participated in only 1 treatment period.) | 2 | 6 | 0 (Participants in Cohort C participated in only 1 treatment period.) | 0 (Participants in Cohort C participated in only 1 treatment period.) | 0 (Participants in Cohort C participated in only 1 treatment period.)
Completed | 0 | 0 | 2 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Placebo: Placebo: once daily (QD) oral dosing for 14 consecutive days
- 35 mg LY2886721: Participants received 35 mg LY2886721: oral dosing for 14 consecutive days
- 70 mg LY2886721: Participants received 70 mg LY2886721: single oral dose followed by QD oral dosing for 14 consecutive days or single oral dose.
- 140 mg LY2886721: Participants received 140 mg LY2886721: single oral dose
- Total: Total of all reporting groups
Arm/Group | Placebo | 35 mg LY2886721 | 70 mg LY2886721 | 140 mg LY2886721 | Total
Number analyzed (Participants) | 8 | 6 | 10 | 6 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 10 | 6 | 30
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 8 | 6 | 10 | 6 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3 | 2 | 8
  Not Hispanic or Latino | 6 | 5 | 7 | 4 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 3 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 2 | 6
  White | 6 | 4 | 5 | 4 | 19
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 6 | 10 | 6 | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant Effects
Description: Data presented are the number of participants who experienced treatment-emergent adverse events. A summary of serious adverse events and other non-serious adverse events, regardless of causality is reported in the Adverse Events module.
Time Frame: Predose up to Day 23
Population: All enrolled participants. Ten participants, 7 in Cohort B and 3 in Cohort C, received 70 mg LY2886721 as a single dose. Six of the participants in Cohort B went on to receive QD dosing for 14 consecutive days. These 6 participants are included in the 70 mg LY2886721 Single Dose arm and the 70 mg LY2886721 Multiple Dose arm.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Placebo: QD oral dosing for 14 consecutive days (Cohort A), single oral dose (Period 1) followed by QD oral dosing for 14 consecutive days (Period 2) (Cohort B), or single oral dose (Cohort C)
- 35 mg LY2886721: 35 mg LY2886721: QD oral dosing for 14 consecutive days (Cohort A)
- 70 mg LY2886721 Multiple Dose: 70 mg LY2886721: single oral dose (Period 1) followed by QD oral dosing for 14 consecutive days (Period 2) (Cohort B)
- 70 mg LY2886721 Single Dose: 70 mg LY2886721: single oral dose (Cohort B [Period 1] and Cohort C)
- 140 mg LY2886721: 140 mg LY2886721: single oral dose (Cohort C)
Arm/Group | Placebo | 35 mg LY2886721 | 70 mg LY2886721 Multiple Dose | 70 mg LY2886721 Single Dose | 140 mg LY2886721
Number analyzed (Participants) | 8 | 6 | 6 | 10 | 6
Participants | 3 | 1 | 3 | 2 | 1

2. Secondary Outcome: Pharmacokinetics: Plasma Maximum Observed Concentration (Cmax) of LY2886721
Time Frame: Day 1 predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours postdose
Population: All randomized participants who received a single 70- or 140-mg dose of LY2886721 and had evaluable single-dose LY2886721 concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | 70 mg LY2886721 Single Dose | 140 mg LY2886721
Number analyzed (Participants) | 10 | 6
nanograms/milliliter (ng/mL) | 182 (26) | 419 (16)

3. Secondary Outcome: Pharmacokinetics: Plasma Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity (AUCinf) of LY2886721
Time Frame: Day 1 predose and 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, and 96 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (ng*hr/mL)
Arm/Group | 70 mg LY2886721 Single Dose | 140 mg LY2886721
Number analyzed (Participants) | 10 | 6
nanograms*hours/milliliter (ng*hr/mL) | 2110 (23) | 4660 (10)

4. Secondary Outcome: Pharmacokinetics: Plasma Maximum Observed Concentration at Steady State (Cmax,ss) of LY2886721
Time Frame: Day 14 predose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours postdose
Population: All randomized participants who received LY2886721 and had evaluable steady-state plasma LY2886721 concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 35 mg LY2886721 | 70 mg LY2886721 Multiple Dose
Number analyzed (Participants) | 6 | 6
ng/mL | 112 (35) | 230 (26)

5. Secondary Outcome: Pharmacokinetics: Plasma Area Under the Concentration Versus Time Curve (AUC) of LY2886721
Description: AUC over the dosing interval at steady state (AUCtau,ss) is reported for participants who received multiple doses of LY2886721.
Time Frame: Day 14 predose and 0.5, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, and 120 hours postdose
Population: All randomized participants who received LY2886721 and had evaluable steady-state plasma LY2886721 concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | 35 mg LY2886721 | 70 mg LY2886721 Multiple Dose
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 1100 (26) | 2400 (24)

6. Secondary Outcome: Percent Change From Baseline in Cerebrospinal Fluid (CSF) Amyloid 1-40 Concentration at Day 15
Description: Least squares (LS) mean percent changes from baseline to Day 15 in CSF amyloid 1-40 concentrations for participants in Cohort B are reported. LS means were calculated from an analysis of covariance (ANCOVA) with treatment group and predose CSF amyloid 1-40 concentration as fixed effects. The 95% confidence interval (CI) of the percent change from baseline was computed by back-transforming the mean difference between endpoint and baseline.
Time Frame: Baseline, Day 15
Population: All randomized participants in Cohort B who received multiple doses of placebo or 70 mg LY2886721 and had evaluable CSF amyloid 1-40 concentrations.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- 70 mg LY2886721 Multiple Dose (Cohort B): 70 mg LY2886721: single oral dose (Period 1) followed by QD oral dosing for 14 consecutive days (Period 2)
Arm/Group | Placebo (Cohort B) | 70 mg LY2886721 Multiple Dose (Cohort B)
Number analyzed (Participants) | 2 | 6
Percent change | -0.97 [-5.81 to 3.87] | -74.46 [-77.25 to -71.67]

7. Secondary Outcome: Percent Change From Baseline in Cerebrospinal Fluid (CSF) Amyloid 1-40 Concentration at 24 Hours Post-dose
Description: LS mean percent changes from baseline to 24 hours post-dose in CSF amyloid 1-40 concentrations for participants in Cohort C are reported. LS means were calculated from an ANCOVA with treatment group and predose CSF amyloid 1-40 concentration as fixed effects. The 95% CI of the percent change from baseline was computed by back-transforming the mean difference between endpoint and baseline.
Time Frame: Baseline, 24 hours post-dose
Population: All randomized participants in Cohort C who received placebo or LY2886721 and had measurable CSF amyloid 1-40 concentration data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Placebo (Cohort C) | 70 mg LY2886721 (Cohort C) | 140 mg LY2886721 (Cohort C)
Number analyzed (Participants) | 3 | 3 | 6
Percent change | -11.59 [-24.50 to 1.32] | -64.75 [-76.38 to -53.13] | -72.05 [-80.36 to -63.74]

ADVERSE EVENTS:
Groups:
- 70 mg LY2886721 Single Dose: 70 mg LY2886721: single oral dose(Cohort B [Period 1] and Cohort C)
Arm/Group | Placebo | 35 mg LY2886721 | 70 mg LY2886721 Multiple Dose | 70 mg LY2886721 Single Dose | 140 mg LY2886721
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/10 | 0/6
Other Adverse Events (participants affected / at risk) | 3/8 | 1/6 | 3/6 | 2/10 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | 35 mg LY2886721 (N=6) | 70 mg LY2886721 Multiple Dose (N=6) | 70 mg LY2886721 Single Dose (N=10) | 140 mg LY2886721 (N=6)
Scotoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural dizziness (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days